CLINICAL TRIAL: NCT04600752
Title: A Multicenter, Open-label, Non-comparative Phase IV Clinical Study to Evaluate the Safety and Clinical Efficacy of Augmentin Extra Strength (ES)-600 in Children With Acute Otitis Media (AOM) in India
Brief Title: Study to Evaluate the Safety and Clinical Efficacy of Augmentin® Extra Strength-600 in Children With Acute Otitis Media in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213514
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-05

CONDITIONS: Otitis Media; Infections, Respiratory Tract; Respiratory Tract Infections
Keywords: Acute otitis media; Augmentin Extra Strength; Amoxicillin-clavulanic acid; Pediatric; Beta-lactamase
MeSH Terms: conditions — Otitis Media; Respiratory Tract Infections | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Intervention Model Description: This is a single arm, multicenter, non-comparative study.
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving Augmentin (ES)-600 (Experimental): Eligible participants will receive Augmentin (ES)-600 at 90/6.4 mg/kg/day administered in two divided doses, every 12 hours with food for 10 days.
  Interventions: Drug: Augmentin (ES)-600

INTERVENTIONS:
Drug: Augmentin (ES)-600 — Augmentin ES will be administered as reconstituted oral suspension containing Amoxicillin and Potassium Clavulanate 600 mg/42.9 mg per 5 milliliters.

SUMMARY:
Augmentin (ES)-600 is a high-dose amoxicillin/clavulanic acid 14:1 formulation that allows administration at 90/6.4 milligrams (mg)/kilograms (kg)/day in two divided doses. Most physicians in India use the standard Augmentin (amoxicillin:clavulanic acid 7:1) (45/6.4 mg/kg/day) formulation and double the dose to achieve higher dose of amoxicillin/clavulanic acid at 90 mg/kg/day in pediatric acute otitis media (AOM) due to non-availability of Augmentin (ES)-600. Using the 7:1 formulation causes unnecessary exposure to higher proportionate dose of clavulanic acid (12.8 mg/kg/day) as a unit dose of 6.4 mg/kg/day of clavulanic acid is only required for efficacy against beta-lactamase producing AOM pathogens. Hence, there is an unmet need for availability of Augmentin (ES)-600 in India. This is an open label, single arm, multicenter, non-comparative study in participants aged 6 months to 12 years with AOM. It aims to assess the safety and clinical efficacy of Augmentin (ES)-600 administered in two divided doses, every 12 hours in pediatric population in India. AUGMENTIN is a registered trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged: 6 months to 12 years; no gender restriction.
* Diagnosis of AOM on basis of otoscopic findings as defined below:

  1. Purulent otorrhea of less than 24 hours duration or
  2. Middle ear effusion
* Middle ear effusion is evidenced by at least two of the following:

  1. Decreased or absent tympanic mobility measured by pneumatic otoscopy,
  2. Yellow or white discoloration of the tympanic membrane, or
  3. Opacification of the tympanic membrane plus

At least one of the following indicators of acute inflammation:

1. Ear pain within 24 hours, including unaccustomed tugging or rubbing of ear,
2. Marked redness of the tympanic membrane, or
3. Distinct fullness or bulging of the tympanic membrane.

   * The participant and parent(s)/legal guardian(s) are willing and able to comply with the study protocol.
   * In accordance with regional/local laws and regulations, the parent(s)/legal guardian(s) has given signed informed, dated consent; and the participant has given written assent, if applicable, to participate in the study.

Exclusion Criteria:

* Weight more than 40 kg.
* Spontaneous perforation of the tympanic membrane and drainage for longer than 24 hours.
* Tympanoplastic tube(s) in place, or has anatomic abnormalities associated with recurrent AOM, prolonged middle ear effusion, including cleft palate or repair, high-arched palate or Down's syndrome.
* A serious underlying disease as per clinician's judgment.
* Concomitant infection which would preclude evaluation of the response of his/her acute otitis media to the study intervention.
* Pre-existing renal insufficiency (plasma creatinine greater than [>]1.5 times upper limit of normal range for age).
* Pre-existing liver disease(s) and/or hepatic dysfunction.
* Evidence of leukopenia and/or thrombocytopenia.
* History of previous hypersensitivity reaction to penicillins, cephalosporins or other beta-lactam antibiotics.
* History of Augmentin-associated cholestatic jaundice/hepatic dysfunction.
* History of phenylketonuria or a known hypersensitivity to aspartame.
* Received, within 48 hours of study entry, or is scheduled to receive during the study period, any medication which may alter bowel function.
* Currently receiving or has received more than one dose of systemic antibiotic therapy within one week prior to the initiation of the study. AOM treatment failures with Amoxicillin, erythromycin, sulfamethoxazole or Trimethoprim-Sulfamethoxazole are not subject to this criterion.
* Receipt of an investigational compound (non-Food and Drug Administration [FDA] and non- Drugs Controller General Of India [DCGI] approved) or device within the previous 30 days or five half-lives, whichever is longer, preceding the first dose of study intervention or during the study.
* Participants with symptoms suggestive of active Coronavirus Disease 2019 (COVID-19) infection (fever, cough, etc).
* Participants with known COVID-19 positive contacts within the past 14 days.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-11-12 (Actual); Study Completion 2022-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- India (13):
  - GSK Investigational Site, Raipur, Chhattisgarh
  - GSK Investigational Site, Jaipur, Rajasthan
  - GSK Investigational Site, Varanasi, Uttar Pradesh
  - GSK Investigational Site, Belgaun
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Kanpur
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Ludhiana
  - GSK Investigational Site, Madurai
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Purne

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was an open label, multicenter, non-comparative study. Participants were children aged between 6 months to 12 years, presenting with Acute respiratory tract infections (ARTIs) including Acute otitis media (AOM), Acute bacterial rhinosinusitis (ABRS) and Community acquired bacterial pneumonia (CABP)
Groups:
- Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600: Participants with AOM were administered with Augmentin Extra Strength (ES)-600 at 90/6.4 milligram (mg)/ kilogram (kg)/day administered in two equally divided doses, 12 hours apart with food for 10 days. The formulation Augmentin (ES)-600 is Amoxicillin and potassium clavulanate oral suspension IP 600 mg/42.9 mg per 5 milliliter (mL)
- Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600: Participants with ABRS were administered with Augmentin (ES)-600 at 90/6.4 mg/kg/day administered in two equally divided doses, 12 hours apart with food for 10 days. The formulation Augmentin (ES)-600 is Amoxicillin and potassium clavulanate oral suspension IP 600 mg/42.9 mg per 5 milliliter (mL)
- Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600: Participants with CABP were administered with Augmentin (ES)-600 at 90/6.4 mg/kg/day administered in two equally divided doses, 12 hours apart with food for 10 days. The formulation Augmentin (ES)-600 is Amoxicillin and potassium clavulanate oral suspension IP 600 mg/42.9 mg per 5 milliliter (mL)
Period: Overall Study
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
Started | 136 | 106 | 68
Completed | 133 | 104 | 67
Not Completed | 3 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600 | Total
Number analyzed (Participants) | 136 | 106 | 68 | 310
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.869 (2.9995) | 4.404 (3.0134) | 2.592 (2.0324) | 3.772 (2.8913)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 39 | 16 | 115
  Male | 76 | 67 | 52 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 136 | 106 | 68 | 310
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 136 | 106 | 68 | 310

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A treatment emergent AE event has its onset date on or after treatment start date and on or before treatment stop date + 1 day
Time Frame: Up to 28 days
Population: Intent to Treat Population (ITT) which included all participants who are enrolled and received at least 1 dose of Augmentin (ES)-600.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
Number analyzed (Participants) | 136 | 106 | 68
Participants | 10 | 3 | 3

2. Secondary Outcome: Number of Participants With Early Clinical Response at On-therapy (OT) Visit
Description: Early clinical response was categorized as treatment 'success' or treatment 'failure' at OT Visit (Day 3 to 5). Success was defined as 'clinical cure' that included sufficient resolution or improvement of the signs and symptoms such that no additional antibiotic therapy was indicated or 'improvement' that included improvement in at least 1 presenting signs/symptoms such that no additional antibiotic indicated. Failure is defined as 'Clinical Failure' that included as non-improvement or deterioration in any sign/symptoms after 2 or more days of therapy and additional antibiotic therapy is indicated or 'Unable to Determine' included a valid assessment of clinical outcome could not be made (eg, participant did not attend or consent to clinical examination or lost to follow-up). Participants who were not taking minimum 4 doses in two days were categorized as non evaluable.
Time Frame: On-therapy (OT) visit (Day 3 to 5)
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
Number analyzed (Participants) | 136 | 106 | 68
Participants
  Success | 134 | 104 | 68
  Failure | 1 | 0 | 0
  Non Evaluable | 1 | 2 | 0

3. Secondary Outcome: Number of Participants With Primary Clinical Response at End of Therapy (EOT)
Description: Primary clinical response at the end-of-therapy visit was categorized as treatment 'success' or treatment 'failure'. Success was defined as 'Clinical Cure' that included sufficient resolution or improvement of the signs and symptoms that no additional antibiotic therapy was indicated or 'Improvement' that included improvement, but incomplete resolution of presenting signs/symptoms and no additional antibiotic indicated. Failure is defined as 'Clinical Failure' that included non-improvement or deterioration in any sign/symptoms after 2 or more days of therapy and additional antibiotic therapy indicated, or 'Unable to determine' defined as a valid assessment of clinical outcome could not be made (e.g., participant did not attend or consent to clinical examination or lost to follow-up). Non-Evaluable is defined as participants who had less than (<) 80% compliance
Time Frame: End of therapy visit (Day 12 to 14)
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
Number analyzed (Participants) | 136 | 106 | 68
Participants
  Success | 132 | 104 | 67
  Failure | 2 | 0 | 1
  Non Evaluable | 2 | 2 | 0

4. Secondary Outcome: Number of Participants With Secondary Clinical Response at Follow-up (FU)
Description: Secondary clinical response at follow-up was categorized as treatment 'success' or treatment 'failure'. Success was defined as 'Persistent clinical cure' that included sufficient resolution of signs/symptoms for those participants who were clinically cured or improved at the end of therapy and no additional antibiotic indicated. Failure was defined as 'Clinical recurrence' that included reappearance of signs/symptoms for those participants who were clinically cured or improved at the end of therapy and additional antibiotic therapy was indicated, or 'Unable to determine' that included valid assessment of clinical outcome could not be made (e.g., participant did not attend end of therapy visit, or extenuating circumstances or lost to follow-up). Participant with missing responses were categorized as 'Missing'.
Time Frame: Follow up visit (Day 22 to 28)
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
Number analyzed (Participants) | 136 | 106 | 68
Participants
  Success | 130 | 104 | 66
  Failure | 0 | 0 | 1
  Missing | 6 | 2 | 1

5. Secondary Outcome: Number of Participants With Protocol-defined Diarrhea (PDD) (Due to Study Medication)
Description: Protocol-defined diarrhea was defined as a) 3 or more watery stools in one day or b) 4 or more loose/watery stools in one day or c) 2 watery stools per day for two consecutive days or d) 3 loose/watery stools per day for two consecutive days.
Time Frame: From OT visit (Day 3 to 5) to FU visit (Day 22-28)
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
Number analyzed (Participants) | 136 | 106 | 68
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All Cause Mortality, Serious Adverse events and Non Serious Adverse events were collected from visit 1 (Day 1) up to follow-up visit (Day 22 to 28)
Description: Intent to Treat Population (ITT) which included all participants who are enrolled and received at least 1 dose of Augmentin (ES)-600
Arm/Group | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/106 | 0/68
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/106 | 0/68
Other Adverse Events (participants affected / at risk) | 10/136 | 3/106 | 3/68
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Acute Otitis Media (AOM) Receiving Augmentin (ES)-600 (N=136) | Participants With Acute Bacterial Rhinosinusitis (ABRS) Receiving Augmentin (ES)-600 (N=106) | Participants With Community Acquired Bacterial Pneumonia (CABP) Receiving Augmentin (ES)-600 (N=68)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (5) | 1 (1) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/52/NCT04600752/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/52/NCT04600752/SAP_001.pdf